CLINICAL TRIAL: NCT03930355
Title: Effect of Perioperative Transfusion on Early and Late Outcome After Major Elective Surgery
Brief Title: Perioperative Transfusion Related Outcome
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Assoc Prof, Diskapi Teaching and Research Hospital
Other Study IDs: TULIP TS II
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-06

CONDITIONS: Blood Transfusion
Keywords: Surgery; Perioperative; Transfusion; Mortality
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfused: Patients who received blood transfusion in the perioperative period
  Interventions: Other: Blood transfusion
- Non transfused: Patients who did not receive blood transfusion in the perioperative period
  Interventions: Other: Control

INTERVENTIONS:
Other: Blood transfusion — Patients who received blood transfusion in the perioperative period
  Groups: Transfused
Other: Control — Patients who did not receive blood transfusion in the perioperative period
  Groups: Non transfused

SUMMARY:
A secondary analysis of the Turkish National Perioperative Transfusion Study (TULIP TS) database will be performed.

DETAILED DESCRIPTION:
The Turkish National Perioperative Transfusion Study (TULIP TS) was conducted by The Turkish Society of Anesthesiologists' Multicentre Clinical Trials Network.

TULIP TS included 6481 patients undergoing major elective surgery, from 61 study sites across the country.

Transfusion practices of clinicians working at diverse surgical fields; differences between current transfusion practices and patient blood management strategies; the areas for improvement and the obstacles that could prevent change were evaluated and identified.

Data relevant to perioperative transfusion rates of red blood cells, fresh frozen plasma and platelets, the indications for transfusion and postoperative adverse outcomes including 1 month all cause mortality was obtained.

The TULIP TS group aims to collect further data concerning 1 year all cause mortality of the same patient population and to evaluate adverse outcomes in transfused and non transfused patients.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing major elective surgery

Exclusion Criteria:

• Trauma patients, emergency surgery

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing major elective surgery in General surgery Orthopedics Urology Transplantation surgery Neurosurgery Gynecology and obstetrics Cardiovascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 6121 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
1 year all cause mortality | postoperative 366th day
  Number of participants died: all cause mortality
Acute kidney injury | postoperative 30th day
  Number of participants with acute kidney injury
Acute respiratory failure | postoperative 30th day
  Number of participants with acute respiratory failure
Thromboembolic event | postoperative 30th day
  Number of participants with a thromboembolic event
Ischemic event | postoperative 30th day
  Number of participants with an ischemic event
Infection | postoperative 30th day
  Number of participants with infection
Myocardial infarction | postoperative 30th day
  Number of participants with myocardial infarction
Adverse cardiac event | postoperative 30th day
  Number of participants with an adverse cardiac event

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ünal, Principal Investigator — Ministry of Health
Locations (60):
- Turkey (Türkiye) (60):
  - Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara
  - Acibadem University Mehmet Ali Aydinlar Atakent Hospital, Ankara
  - Ankara University Cebeci Medical Center, Ankara
  - Ankara University Ibni Sina Hospital, Ankara
  - Başkent University Ankara Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Private Cankaya Hospital, Ankara
  - Ufuk University Medical Faculty Dr. Ridvan Ege Training and Research Hospital, Ankara
  - University of Health sciences Ankara Child Health and Diseases Hematology Oncology Training and research Hospital, Ankara
  - University of Health Sciences Ankara Numune Training and Research Hospital, Ankara
  - University of Health Sciences Ankara Training and Research Hospital, Ankara
  - University of Health Sciences Diskapi Yildirim Beyazit Trainig Research Hospital, Ankara
  - University of Health Sciences Dr Abdurrahman Yurtaslanı Ankara Oncology Training and Research Hospital, Ankara
  - University of Health Sciences Kecioren Training and Research Hospital, Ankara
  - University of Health Sciences Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara
  - University of Health Sciences Yenimahalle Training and Research Hospital, Ankara
  - University of Health Sciences Zubeyde Hanim Gynecology and Maternity Training and Research Hospital, Ankara
  - University of Technology and Economics Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - University of Health Sciences Antalya Training and Research Hospital, Antalya
  - Balikesir University Training and Research Hospital, Balıkesir
  - Uludağ University Medical Faculty, Bursa
  - University of Health Sciences Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Hitit University Corum Erol Olcok Training and Research Hospital, Çorum
  - Trakya University Medical Faculty, Edirne
  - Fırat University Medical Faculty, Elâzığ
  - Erzincan University Mengucek Gazi Training and Research Hospital, Erzincan
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir
  - Suleyman Demirel University Medical Faculty, Isparta
  - Acibadem University Altunizade Hospital, Istanbul
  - Istanbul University Medical Faculty, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - University of Health Sciences Fatih Sultan Mehmet Training and Research Hospital, Istanbul
  - University of Health Sciences Haydarpasa Numne Training and Research Hospital, Istanbul
  - University of Health Sciences Istanbul Training and Research Hospital, Istanbul
  - University of Health Sciences Kanuni Sultan Suleyman Training and Research Hospital, Istanbul
  - University of Health Sciences Okmeydanı Training and Research Hospital, Istanbul
  - University of Health Sciences Umraniye Training and Research Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - University of Health Sciences Bozyaka Training Research Hospital, Izmir
  - University of Health Sciences İzmir Tepecik Training and Research Hospital, Izmir
  - Sutcu Imam University Medical Faculty, Kahramanmaraş
  - Erciyes University Medical Faculty, Kayseri
  - Anadolu Health Center Hospital, Kocaeli
  - University of Health Sciences Derince Training and Research Hospital, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty Center for Health and Research, Konya
  - Selcuk University Medical Faculty, Konya
  - University of Health Sciences Konya Training and Research Hospital, Konya
  - Inonu University Liver Transplantation Institute, Malatya
  - Manisa Celal Bayar University Medical Faculty Hafsa Sultan Hospital, Manisa
  - Mersin University Medical Faculty, Mersin
  - Ordu University Medical Faculty, Ordu
  - Osmaniye State Hospital, Osmaniye
  - Ondokuz Mayıs University Medical Faculty, Samsun
  - Namık Kemal University Medical Faculty, Tekirdağ
  - Karadeniz Technical University Medical Faculty Farabi Hospital, Trabzon
  - Tunceli State Hospital, Tunceli
  - Van Yuzuncuyıl University Medical Faculty Dursun Odabası Center, Van
  - Bulent Ecevit University Medical Faculty Center for Health and Research, Zonguldak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meier J, Filipescu D, Kozek-Langenecker S, Llau Pitarch J, Mallett S, Martus P, Matot I; ETPOS collaborators. Intraoperative transfusion practices in Europe. Br J Anaesth. 2016 Feb;116(2):255-61. doi: 10.1093/bja/aev456. PMID 26787795
- [Background] Kalil AC, Mattei J, Florescu DF, Sun J, Kalil RS. Recommendations for the assessment and reporting of multivariable logistic regression in transplantation literature. Am J Transplant. 2010 Jul;10(7):1686-94. doi: 10.1111/j.1600-6143.2010.03141.x. PMID 20642690
- [Result] Kotze A, Carter LA, Scally AJ. Effect of a patient blood management programme on preoperative anaemia, transfusion rate, and outcome after primary hip or knee arthroplasty: a quality improvement cycle. Br J Anaesth. 2012 Jun;108(6):943-52. doi: 10.1093/bja/aes135. PMID 22593128
- [Result] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460